CLINICAL TRIAL: NCT02963480
Title: Investigation of Inflammatory Parameters in a Perioperative Closed-meshed Standard Progress in CPB Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Martin Bernardi, Dr., Medical University of Vienna
Other Study IDs: 1518/2016
Record Dates: First submitted 2016-07-06; First posted 2016-11-15 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis: Patients, who developed postoperative sepsis
  Interventions: Procedure: Cardiac Surgery
- SIRS: Patients, who developed postoperative SIRS
  Interventions: Procedure: Cardiac Surgery

INTERVENTIONS:
Procedure: Cardiac Surgery

SUMMARY:
Similar to poly-trauma, acute myocardial infarction, or stroke, the speed and appropriateness of therapy administered in the initial hours after severe sepsis develops are likely to influence outcome. However, the crux of matter is the "early diagnosis" lacking of high sensitive and specific test, in contrary to, for instance, the acute coronary syndrome, where the highly sensitive Troponin T is measured and increased values are fix component of the diagnosis and definition of acute myocardial infarction. Cardiac surgery can initiate a systemic inflammatory response syndrome (SIRS) induced by extrinsic and intrinsic factors, which are associated in the pathogenesis of postoperative complications. SIRS is closely related to sepsis, but in contrast sepsis is induced by infection. This strong inflammatory response induces malfunction of the peripheral circulation with increased lactate levels, pronounced fluid accumulation and increased need of vasopressors.

The investigators want to assess the timing dynamic of release of IL-6 apart from established markers like CRP, leukocytes, PCT. Target of this is to estimate the time-scope and -advance of an "IL-6 axis panel" toward the measurement of standard inflammation parameters in inflammatory response to surgical trauma as a pre-figuration of non-infectious SIRS and to search for a eligible "cut-off" of IL-6.

DETAILED DESCRIPTION:
Similarly for early detection of SIRS/Sepsis, interleukin 6 (IL-6) assays have been brought up for discussion and have been studied extensively over last years. IL-6 is pro-and anti-inflammatory cytokine with multimodal functions in physiology and patho- physiology: As a major regulator of hepatic acute phase response, IL-6 induces the expression of C- reactive protein, fibrinogen and serum amyloid-A protein among others. However, along with pro-inflammatory effects IL-6 is described as an anti- inflammatory agent. Especially in systemic inflammatory response syndrome (SIRS) and sepsis the pro-inflammatory impact of IL-6 is of paramount interest: Via trans-signaling using the soluble IL-6 receptor (sIL-6R) pathway adherent junctions of endothelial VE-cadherin are disconnected causing a loss of barrier function. Increased endothelial permeability results in trans-endothelial flow of fluid and interstitial oedema with consecutive impairment of tissue oxygenation and increased blood viscosity.

Recent publications suggest, that regenerative or anti-inflammatory activities of IL-6 are mediated by classic signalling via a membrane bound IL-6 receptor, whereas pro-inflammatory responses of interleukin-6 are rather mediated by trans-signalling using soluble IL-6.

The IL-6, sIL-6R, soluble glycoprotein 130- buffer:

Since all cells in body express glycoprotein (gp) 130, one of the crucial molecules in signal-transduction of IL-6, they all are susceptible to activation by the complex of IL-6 and sIL-6-Receptor. Thus, under steady state conditions there must be a control mechanism, which prevents IL-6/sIL-6R trans-signalling and hence unbounded activation of pro- inflammatory axis conterminously with a kind of "buffer system" for the IL-6 activity. For such a buffer, at least three different molecules have been taken into account: IL-6 itself, the -above mentioned- sIL-6Receptor and the soluble form of gp130 (sgp130).

Under steady-state and non- inflammatory conditions levels of sIL-6R and sgp130 are almost 1000 fold higher than IL-6, meaning IL-6 is once secreted, it will form a complex with sIL-6R and consecutively will be neutralized by association to sgp130. The immunological impact of circulating IL-6 is a function of the serum IL-6, sIL-6R and sgp130 concentration, respectively of the proportion of the proteins to each other.

Kinetic of IL-6 and the impact of procalcitonin:

In the early nineties, the use of procalcitonin (PCT) has been described by Assicot et al. for the diagnosis of, in particular, bacterial sepsis. However, for discrimination of the acute inflammatory pattern of sepsis from other causes of generalized inflammation (e.g., postoperative, other forms of shock) no recommendation has been given for the use PCT to distinguish between severe infection and other acute inflammatory states in the actual guidelines. Nevertheless, conflicting to this reference, a recent high impact meta-analysis concluded that PCT can differentiate effectively between sepsis and systemic inflammatory response syndrome (SIRS) of non- infectious origin with a cut-off of between 1·0 and 2·0 ng/mL.

The drawback of PCT and e.g. C-reactive Protein (CRP) in relation to members of the IL-6 axis is, that these molecules are downstream of the IL-6 axis and therefore the increase caused by endotoxin or for instance by surgical trauma is delayed.

ELIGIBILITY:
Exclusion Criteria:

* Emergency procedures
* Heart transplantation
* Elective left ventricular assist device (LVAD) implantation
* Pulmonary thrombendarterectomy
* Declined informed consent
* Chronic renal failure on renal replacement therapy
* Body mass index < 18
* Age < 18 years
* Pregnant woman
* Receiving chemotherapy or diagnosed with any disease state (e.g., AIDS)

that has produced leukopenia

* Receiving anti-leucocyte drugs, immunosuppression or TNF-α Blockers
* CRP > 2mg.dl-1
* Patients receiving postoperative extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational cohort study in patients with elective cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change of IL-6 | 10 days
  Change of IL-6 over the observation period, peak and nadir comparison

SECONDARY OUTCOMES:
Change of PCT | 10 days
  Change of PCT over the observation period, peak and nadir comparison
Change of bioelectrical impedance analysis | 10 days
  Change of percent Total Body Water, Fat Free Mass over the observation period

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Bernardi, MD, Principal Investigator — Medical University of Vienna, Dept. of Cardiothoracic and Vascular Anesthesia and Intensive Care
Locations (1):
- Divison of Cardiothoracic Anaesthesia and Intensive Care, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Marshall JC, Reinhart K; International Sepsis Forum. Biomarkers of sepsis. Crit Care Med. 2009 Jul;37(7):2290-8. doi: 10.1097/CCM.0b013e3181a02afc. PMID 19487943
- [Background] Alpert JS, Thygesen K, Antman E, Bassand JP. Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. J Am Coll Cardiol. 2000 Sep;36(3):959-69. doi: 10.1016/s0735-1097(00)00804-4. PMID 10987628
- [Background] Bernardi MH, Rinoesl H, Dragosits K, Ristl R, Hoffelner F, Opfermann P, Lamm C, Preissing F, Wiedemann D, Hiesmayr MJ, Spittler A. Effect of hemoadsorption during cardiopulmonary bypass surgery - a blinded, randomized, controlled pilot study using a novel adsorbent. Crit Care. 2016 Apr 9;20:96. doi: 10.1186/s13054-016-1270-0. PMID 27059056
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Evans BJ, Haskard DO, Finch JR, Hambleton IR, Landis RC, Taylor KM. The inflammatory effect of cardiopulmonary bypass on leukocyte extravasation in vivo. J Thorac Cardiovasc Surg. 2008 May;135(5):999-1006. doi: 10.1016/j.jtcvs.2007.08.071. PMID 18455576
- [Background] Chalaris A, Garbers C, Rabe B, Rose-John S, Scheller J. The soluble Interleukin 6 receptor: generation and role in inflammation and cancer. Eur J Cell Biol. 2011 Jun-Jul;90(6-7):484-94. doi: 10.1016/j.ejcb.2010.10.007. Epub 2010 Dec 8. PMID 21145125
- [Background] Wolsk E, Mygind H, Grondahl TS, Pedersen BK, van Hall G. IL-6 selectively stimulates fat metabolism in human skeletal muscle. Am J Physiol Endocrinol Metab. 2010 Nov;299(5):E832-40. doi: 10.1152/ajpendo.00328.2010. Epub 2010 Sep 7. PMID 20823453
- [Background] Kruttgen A, Rose-John S. Interleukin-6 in sepsis and capillary leakage syndrome. J Interferon Cytokine Res. 2012 Feb;32(2):60-5. doi: 10.1089/jir.2011.0062. Epub 2011 Dec 2. PMID 22136372
- [Background] Scheller J, Chalaris A, Schmidt-Arras D, Rose-John S. The pro- and anti-inflammatory properties of the cytokine interleukin-6. Biochim Biophys Acta. 2011 May;1813(5):878-88. doi: 10.1016/j.bbamcr.2011.01.034. Epub 2011 Feb 4. PMID 21296109
- [Background] Jones SA, Scheller J, Rose-John S. Therapeutic strategies for the clinical blockade of IL-6/gp130 signaling. J Clin Invest. 2011 Sep;121(9):3375-83. doi: 10.1172/JCI57158. Epub 2011 Sep 1. PMID 21881215
- [Background] Rose-John S. IL-6 trans-signaling via the soluble IL-6 receptor: importance for the pro-inflammatory activities of IL-6. Int J Biol Sci. 2012;8(9):1237-47. doi: 10.7150/ijbs.4989. Epub 2012 Oct 24. PMID 23136552
- [Background] Assicot M, Gendrel D, Carsin H, Raymond J, Guilbaud J, Bohuon C. High serum procalcitonin concentrations in patients with sepsis and infection. Lancet. 1993 Feb 27;341(8844):515-8. doi: 10.1016/0140-6736(93)90277-n. PMID 8094770
- [Background] Wacker C, Prkno A, Brunkhorst FM, Schlattmann P. Procalcitonin as a diagnostic marker for sepsis: a systematic review and meta-analysis. Lancet Infect Dis. 2013 May;13(5):426-35. doi: 10.1016/S1473-3099(12)70323-7. Epub 2013 Feb 1. PMID 23375419